CLINICAL TRIAL: NCT06208449
Title: Comparison of Robotic Versus Thoracoscopy Versus Thoracotomy Repair for Congenital Esophageal Atresia
Brief Title: Robotic Versus Thoracoscopy Versus Thoracotomy Repair for Congenital Esophageal Atresia
Acronym: RR VS TR VS OR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zunyi Medical College (Other)
Collaborators: Guiyang Children's Hospital (Unknown); Guizhou Provincial People's Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Binzhou Medical University (Other)
Responsible Party: Principal Investigator, zebing Zheng, prof., Zunyi Medical College
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: esophageal atresia; 82060100 (Other Grant/Funding Number: National Natural Science Foundation of China); ZK-2021-361 (Other Grant/Funding Number: Basic Research Project of Guizhou Province)
Record Dates: First submitted 2024-01-01; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Congenital Esophageal Atresia
Keywords: robotic surgery; thoracoscopy repair; thoracotomy repair; esophageal atresia; efficacy; complications
MeSH Terms: conditions — Esophageal Atresia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Robotic repair group (Experimental): 1. the patients were lying in a left decubitus position (45° prone).
  2. An 8-mm trocar was inserted into the thoracic cavity at the fifth intercostal space of the right midaxillary line and used as a camera port, Another two 8-mm trocars were placed at the third intercostal space of the right midaxillary line and the eighth intercostal space of the posterior axillary line. Insufflation of the CO2 was at a flow rate of 1 L/min and a pressure of 6 mm Hg.
  3. The fistula was ligated and sutured by figure-of-eight suture ligation. The proximal blind end was fully mobilized and the distal blind end was properly mobilized to prepare for anastomosis.
  4. Next, the 5-0 absorbable sutures were used to perform the anastomosis posteriorly and anteriorly in an interrupted way.. Thereafter, the nasogastric tube was inserted into the stomach. followed by another 6 sutures to complete the anterior wall anastomosis.
  5. A chest drain was placed alongside the anastomosis.
  Interventions: Procedure: Robotic repair for EA
- Thoracoscopic repair group (Experimental): 1. All procedures were performed through three ports
  2. Insufflation of the CO2 was at a flow rate of 1 L/min and a pressure of 4-6 mm Hg.
  3. The azygos vein was ligated and cut, or divided by electrocoagulation.
  4. The fistula was then dissociated, ligated with 4-0 absorbable sutures, and divided.
  5. After identifying the proximal esophageal pouch with a nasogastatic tube, the proximal and distal blind ends were mobilized to prepare for anastomosis.
  6. Next, the tip of the blind ends was excised, and the anastomosis was completed with 5-0 absorbable sutures in an interrupted manner.
  7. A chest drain was placed alongside the anastomosis.
  Interventions: Procedure: Thoracoscopic repair for EA
- Thoracotomy repair (Active Comparator): Usually, the fifth intercostal space was applied using the muscular-sparing technique. Fistula ligation, proximal pouch isolation and anastomosis were performed in turn.The fistula was then dissociated, ligated with 4-0 absorbable sutures, and divided. After identifying the proximal esophageal pouch with a nasogastatic tube, the proximal and distal blind ends were mobilized to prepare for anastomosis. Next, the tip of the blind ends was excised, and the anastomosis was completed with 5-0 absorbable sutures in an interrupted manner. A chest drain was placed alongside the anastomosis.
  Interventions: Procedure: Thoracotomy repair for EA

INTERVENTIONS:
Procedure: Robotic repair for EA — The paitents with EA were repaired by Da Vinci robot
  Arms: Robotic repair group
Procedure: Thoracoscopic repair for EA — The patients with EA were repaired by thoracoscopy
  Arms: Thoracoscopic repair group
Procedure: Thoracotomy repair for EA — The patients with EA were repaired by traditional open thoracotomy.
  Arms: Thoracotomy repair

SUMMARY:
Thoracotomy repair has long been considered the gold standard for the repair of esophageal atresia but is associated with potential musculoskeletal complications which may result in long term morbidity for the patient. thoracoscopy repair offers better visualization of the posterior mediastinal structures, while limiting the surgical trauma. However, studies have shown that the incidence of anastomotic leakage and anastomotic stricture in thoracoscopic repair is not significantly lower than thoracostomy repair. Robotic repair had shorter anastomotic time, lower incidence of anastomotic leakage and stricture, and lower unplanned readmission rate than the thoracotomy repair. However, there were no randomized controlled trials to verify the effectiveness of three procedures. The objection was to compare the difference between robotic repair and thoracoscopic repair, and thoracotomy repair in intraoperative parameters and postoperative complications in EA neonates.

DETAILED DESCRIPTION:
Esophageal atresia (EA) and tracheoesophageal fistula (TEF) is one of the most common congenital malformations of esophagus, with an incidence of 1/2500~1/4500. The condition can be an isolated malformation or may be associated with other congenital anomalies. Since Dr Cameron Height performed the first successful primary repair of a neonate with EA/ TEF in 1941, many advances in surgical technique and neonatal care have steadily improved survival rates of babies within the EA/TEF spectrum. Survival of infants with esophageal atresia has increased over time since the first successful repair and the overall survival exceeds 90%. Commonly, esophageal atresia is repaired via a right posterolateral thoracotomy and more recently muscle sparing thoracotomy has become an alternative to the traditional muscle cutting approach. Open repair has long been considered the gold standard for the repair of esophageal atresia but is associated with potential musculoskeletal complications which may result in long term morbidity for the patient.

The first successful thoracoscopic surgery of a child with EA was reported in 1999. Compared to thoracotomy repair the proposed main advantage of thoracoscopic repair is that it offers better visualization of the posterior mediastinal structures, while limiting the surgical trauma. However, studies have shown that the incidence of anastomotic leakage and anastomotic stricture in thoracoscopic repair is not significantly lower than thoracostomy repair, thoracoscopic repair also offers concerns with more complicated anesthesia, limited workspace, and difficultly controlling the vascular structures. Especially, suturing within such a small, closed space has been considered a major technical difficulty.

Robotic repair was first reported by Meehan in 2009, followed by several case reports. The reported reasons for conversion mainly focused on the incompatibility between the robotic trocar's size and the intercostal space's width, and the technical challenges due to instrument collisions in the extremely limited thoracoscopic space. The intercostal space of neonates is highly narrow, and the thoracic diameter is only 8 cm. These are the two key technical issues to be addressed in this study. According to the existing robotic system setup standard for adults, the distance required between trocar ports in robots is usually at least 8 cm to ensure sufficient operating space and avoid instrument collisions. Even for the new generation of robots, this minimum distance requires 5-6 cm. Huge robotic trocars used in EA neonates fail to meet the standard for conventional operating port distances. There have study designed an asymmetric port distribution technique in which the third and eighth intercostal ports are 3 cm and 5 cm away from the camera port. The surgeons primarily manipulated the inner-articulating part of the robotic arms within the thoracic cavity, avoiding instrument collisions outside. Moreover, the setup of the trocars ensures that the robotic arms can reach the main operating area. When combined with instruments of 7 degrees of freedom, the mobilization and anastomosis of the esophagus could be completed easily, breaking through the narrow space restriction of thoracic cavity. Inserting 8-12 cm trocars into tiny intercostal space was another technical challenge. The results shown the robotic repair had shorter anastomotic time, lower incidence of anastomotic leakage and stricture, and lower unplanned readmission rate than the thoracotomy repair.

An international survey from 2014 highlighted the need for consensus on the optimal surgical treatment of EA. However, a detailed understanding of whether thoracoscopic repair or robotic repair offers advantages in terms of health outcomes, safety, and efficacy for providers compared to thoracotomy repair is still lacking. Several reviews are opinion-based or obscured by institutional/personal experiences. Herewith, we designed a comprehensive study and focused on evaluating the difference between robotic repair and thoracoscopic repair, and thoracotomy repair in intraoperative parameters and postoperative complications in EA neonates.

ELIGIBILITY:
Inclusion Criteria:

* Type C EA neonates with short esophageal gap length (less than 3 vertebral bodies), mini-invasive repair, and a successful one-stage anastomosis were included.

Exclusion Criteria:

* Patients with respiratory distress requiring assisted ventilation, long esophageal gap length, multistage surgery, other types EA (type A/B/D/E) or surgical contraindications were excluded.

Gestational age less than 35 weeks and birth weight less than 2kg were excluded.

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
anastomotic leak | 1 year
  anastomotic leak within 30-days postoperative
anastomotic stricture | 1 year
  stricture requiring dilation within 1 year

SECONDARY OUTCOMES:
vocal cord paresis/paralysis at discharge | 1 year
  Vocal cord paresis/paralysis was assessed in patients with symptoms such as aspiration or change in cry prompting a bronchoscopy for conﬁrmation.
time to anastomotic stricture | 2 years
  The time from surgery to the first occurrence of esophageal stenosis requiring dilation
number of dilations in 1 year | 1 year
  The number of dilations of esophageal stenosis in 1 year
esophageal dehiscence | 1 year
  The number of esophageal dehiscence happened in intraoperation.
surgical site infection | 1 year
  Infection of surgical incision
sepsis | 2 year
  Including severe pulmonary infections and sepsis caused by pleural effusion
The use of vasopressors | 1 year
  Include the use of preoperative, intraoperative, postoperative vasopressors.
Ventilation time | 1 year
  Include the usage time preoperative and postoperative ventilation.
Time to full enteral feeds | 1 year
  Time to full enteral feeds
Time to extubation | 1 year
  the time to extubation
Postoperative length of stay | 1 year
  Postoperative length of stay
mortality | 1 year
  Include the alive 30-days postoperation and died within 30-days

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated hospital of zunyi medical university, Zunyi, Guizhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang M, Huang J, Jin Z, Zhang X, Zhou Y, Chi S, Rong L, Zhang Y, Cao G, Li S, Tang ST. Comparison of robotic versus thoracoscopic repair for congenital esophageal atresia: a propensity score matching analysis. Int J Surg. 2024 Feb 1;110(2):891-901. doi: 10.1097/JS9.0000000000000889. PMID 37983822
- [Background] Yang S, Wang P, Yang Z, Li S, Liao J, Hua K, Zhang Y, Zhao Y, Gu Y, Li S, Chen Y, Huang J. Clinical comparison between thoracoscopic and thoracotomy repair of Gross type C esophageal atresia. BMC Surg. 2021 Nov 22;21(1):403. doi: 10.1186/s12893-021-01360-7. PMID 34809633
- [Background] Marquart JP, Bowder AN, Bence CM, St Peter SD, Gadepalli SK, Sato TT, Szabo A, Minneci PC, Hirschl RB, Rymeski BA, Downard CD, Markel TA, Deans KJ, Fallat ME, Fraser JD, Grabowski JE, Helmrath MA, Kabre RD, Kohler JE, Landman MP, Lawrence AE, Leys CM, Mak GZ, Port E, Saito J, Silverberg J, Slidell MB, Wright TN, Lal DR; Midwest Pediatric Surgery Consortium. Thoracoscopy versus thoracotomy for esophageal atresia and tracheoesophageal fistula: Outcomes from the Midwest Pediatric Surgery Consortium. J Pediatr Surg. 2023 Jan;58(1):27-33. doi: 10.1016/j.jpedsurg.2022.09.015. Epub 2022 Sep 24. PMID 36283849